CLINICAL TRIAL: NCT00827242
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multinational Study to Evaluate the Efficacy and Safety of Daily Tadalafil for 12 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Study to Treat Patients Who Have Signs and Symptoms of Benign Prostatic Hyperplasia (BPH) With Tadalafil Daily
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10893; H6D-MC-LVHJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Signs and Symptoms; Prostatic Hyperplasia; Hyperplasia; Genital Diseases, Male; Prostatic Diseases; BPH-LUTS
MeSH Terms: conditions — Prostatic Hyperplasia; Signs and Symptoms; Hyperplasia; Genital Diseases, Male; Prostatic Diseases | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tadalafil (Experimental)
  Interventions: Drug: tadalafil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Following a 4-week placebo lead-in period, subjects received placebo tablet by mouth once daily over a 12-week period.
  Arms: Placebo
Drug: tadalafil — Following a 4-week placebo lead-in period, subjects received tadalafil 5 mg tablet by mouth once daily over a 12-week period.
  Other Names: Cialis; LY450190
  Arms: Tadalafil

SUMMARY:
The purpose of this study is to determine whether an experimental drug known as tadalafil given once daily can reduce the symptoms associated with Benign Prostatic Hyperplasia (straining, urinary frequency, feeling like your bladder is still full, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Men 45 years of age or older with Benign Prostatic Hyperplasia (BPH) also referred to as BPH-LUTS [lower urinary tract symptoms] based on the disease diagnostic criteria at the start of study.
* Provide signed informed consent at the start of the study.
* Have not taken Finasteride therapy for at least 3 months before study drug is dispensed and Dutasteride therapy for at least 6 months before study drug is dispensed.
* Have not taken other BPH therapy (including herbal preparations), overactive bladder (OAB) therapy, or erectile dysfunction (ED) therapy for at least 4 weeks prior to study drug is dispensed.
* Agree not to use any other approved or experimental pharmacologic BPH, OAB, or ED treatments anytime during the study
* Have LUTS with a Total International Prostate Symptom Score (IPSS) greater than or equal to 13 when study drug is dispensed.
* Have reduced peak urine flow rate when study drug is dispensed (measured by a special toilet equipment).
* Demonstrate compliance with study drug administration requirements.

Exclusion Criteria:

* Treated with nitrates for a cardiac conditions.
* Have unstable angina or angina that requires treatment.
* Have had any of the following in the past 90 days: Heart attack, also known as a myocardial infarction (MI); Heart bypass surgery (called coronary artery bypass graft surgery); Had a procedure to open up blood vessels in the heart known as angioplasty or stent placement (percutaneous coronary intervention).
* Have very high or very low blood pressure
* Have problems with kidneys, liver, or nervous system.
* Have uncontrolled diabetes.
* Have had a stroke or a significant injury to brain or spinal cord.
* Have prostate cancer, are being treated for cancer or have clinical evidence of prostate cancer (Prostate-Specific Antigen [PSA] greater than 10 nanograms/milliliter [ng/ml] at the start of study).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2009-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntsville, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middlebury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sarasota, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bay Shore, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Williamsville, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Virginia Beach, Virginia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mühlacker
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oranienburg
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orbassano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
- Mexico (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saltillo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zapopan

REFERENCES:
- [Derived] Vlachopoulos C, Oelke M, Maggi M, Mulhall JP, Rosenberg MT, Brock GB, Esler A, Buttner H. Impact of cardiovascular risk factors and related comorbid conditions and medical therapy reported at baseline on the treatment response to tadalafil 5 mg once-daily in men with lower urinary tract symptoms associated with benign prostatic hyperplasia: an integrated analysis of four randomised, double-blind, placebo-controlled, clinical trials. Int J Clin Pract. 2015 Dec;69(12):1496-507. doi: 10.1111/ijcp.12722. Epub 2015 Aug 24. PMID 26299520
- [Derived] Porst H, Kim ED, Casabe AR, Mirone V, Secrest RJ, Xu L, Sundin DP, Viktrup L; LVHJ study team. Efficacy and safety of tadalafil once daily in the treatment of men with lower urinary tract symptoms suggestive of benign prostatic hyperplasia: results of an international randomized, double-blind, placebo-controlled trial. Eur Urol. 2011 Nov;60(5):1105-13. doi: 10.1016/j.eururo.2011.08.005. Epub 2011 Aug 12. PMID 21871706

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil: Following screening, a 4-week washout period (if needed) and a 4-week placebo lead-in period, subjects were randomized to receive tadalafil 5 mg orally once daily over a 12-week period.
- Placebo: Following screening, a 4-week washout period (if needed) and a 4-week placebo lead-in period, subjects were randomized to receive placebo orally once daily over a 12-week period.
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 161 | 164
Completed | 148 | 152
Not Completed | 13 | 12
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 0 | 3
Not completed — Adverse Event Excluding Death | 2 | 1
Not completed — Entry Criteria Not Met | 4 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 161 | 164 | 325
Age Continuous [Mean (Standard Deviation); unit: years] | 65.1 (8.43) | 64.6 (10.03) | 64.9 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 161 | 164 | 325
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 44 | 90
  Not Hispanic or Latino | 115 | 120 | 235
Race (NIH/OMB) [Count of Participants; unit: Participants] — If a subject reported multiple race categories, he was counted as "more than one race", but not in any single category.
  Participants
    American Indian or Alaska Native | 9 | 8 | 17
    Asian | 2 | 0 | 2
    Black or African American | 3 | 5 | 8
    White | 146 | 150 | 296
    More than one race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 52 | 102
  South America | 43 | 43 | 86
  Europe | 68 | 69 | 137
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram (kg)/meter (m)^2] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilogram (kg)/meter (m)^2 | 27.1 (3.82) | 28.4 (4.21) | 27.7 (4.07)
Baseline Lower Urinary Tract Symptoms (LUTS) Severity [Number; unit: participants] — Baseline LUTS severity was assessed using the International Prostate Symptom Score (IPSS). The IPSS Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Moderate was considered an IPSS score <20. Severe was considered an IPSS>=20.
  participants
    Moderate | 100 | 110 | 210
    Severe | 61 | 54 | 115
Peak Urine Flow Rate (Qmax) Category [Number; unit: participants] — Participants were categorized by Qmax: defined as the peak urine flow rate (measured in mL/second using standard calibrated flowmeter). Based on measurements from 305 randomized participants with a valid uroflowmetry assessment. Uroflowmetry assessments were considered valid and the data were included in statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 mL to <=550 mL and the volume of voided urine (Vcomp) was >=125 mL.
  participants
    <10 mL/sec | 54 | 62 | 116
    10-15 mL/sec | 78 | 67 | 145
    >15 mL/sec | 20 | 24 | 44
Post-void Residual Volume (PVR) [Mean (Standard Deviation); unit: mL] — The amount of urine remaining in the bladder after void completion.
  mL | 44.9 (44.87) | 63.3 (59.88) | 54.2 (53.70)
Prostate-Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] — PSA is a tumor marker associated with prostate cancer. The participant population includes all randomized subjects with non-missing data (n=164 for placebo and n=160 for tadalafil).
  ng/mL | 2.0 (1.75) | 2.2 (1.72) | 2.1 (1.74)
Erectile Dysfunction (ED) [Number; unit: participants] — ED is defined as a consistent change in the quality of erection adversely affecting subject satisfaction with sexual intercourse.
  participants
    Yes | 112 | 112 | 224
    No | 49 | 52 | 101
ED Severity [Number; unit: participants] — ED is defined as a consistent change in the quality of erection adversely affecting subject satisfaction with sexual intercourse. Severity is based on investigator's opinion. Participant population includes all randomized subjects with ED.
  participants
    Mild | 34 | 40 | 74
    Moderate | 61 | 59 | 120
    Severe | 17 | 13 | 30
ED Duration [Number; unit: participants] — ED is defined as a consistent change in the quality of erection adversely affecting subject satisfaction with sexual intercourse. Participant population includes all randomized subjects with ED.
  participants
    <1 year | 14 | 17 | 31
    >=1 year | 98 | 95 | 193
Sexually Active with a Female Partner [Number; unit: participants]
  Yes | 128 | 129 | 257
  No | 33 | 35 | 68
Expect to Remain Sexually Active [Number; unit: participants] — Participant population is based on number of randomized subjects who are reported to be sexually active with a female partner.
  participants
    Yes | 127 | 129 | 256
    No | 1 | 0 | 1
Patient Global Impression of Severity (PGI-S) [Number; unit: participants] — Measures patient's perception of severity of illness at the time of assessment. The responses were grouped into an ordinal scale with 4 categories: normal; mild; moderate; and severe, and were based on postponing urination, straining to begin urination, a weak urinary stream, stopping and restarting urination several times when urinating, prolonged urination with the end of urine flow slowing to a trickle, bladder not feeling emptied after urinating, having to urinate again less than two hours after the last time urinating, accidental urinary leakage, or having to get up at night to urinate.
  participants
    Normal | 5 | 8 | 13
    Mild | 35 | 27 | 62
    Moderate | 102 | 105 | 207
    Severe | 19 | 24 | 43
Clinician Global Impression of Severity (CGI-S) [Number; unit: participants] — Measures clinician's perception of severity of illness at the time of assessment. The responses were grouped into an ordinal scale with 4 categories: normal; mild; moderate; and severe, and were based on postponing urination, straining to begin urination, a weak urinary stream, stopping and restarting urination several times when urinating, prolonged urination with the end of urine flow slowing to a trickle, bladder not feeling emptied after urinating, having to urinate again less than two hours after the last time urinating, accidental urinary leakage, or having to get up at night to urinate.
  participants
    Normal | 0 | 1 | 1
    Mild | 36 | 37 | 73
    Moderate | 104 | 95 | 199
    Severe | 21 | 31 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Weeks, International Prostate Symptom Score (IPSS)
Description: The IPSS Total Score is obtained by combining the scores of the responses to Question 1 through Question 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. Least squares (LS) mean of change from baseline to endpoint is from an analysis of covariance (ANCOVA). The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population was defined as all subjects who were randomized, started study medication, and had non-missing data at baseline and at least one post-baseline visit. The Last Observation Carried Forward (LOCF) imputation technique was employed.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 164
Units on a Scale | -5.6 (0.47) | -3.6 (0.47)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.004, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IPSS. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -1.9, Standard Error of Mean 0.66

2. Secondary Outcome: Change From Baseline to 4 Weeks, Benign Prostatic Hyperplasia (BPH) Impact Index
Description: The BPH Impact Index (BII) is a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores range from 0 to 13; higher scores represent increased perceived impact of benign prostatic hyperplasia-lower urinary tract symptoms on overall health. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 4 weeks
Population: The analysis population includes all subjects who were randomized, started study medication, and had non-missing data at baseline and Week 4.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 158 | 162
Units on a Scale | -1.8 (0.18) | -1.2 (0.18)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.029, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 4 weeks between treatment groups for BII. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.26

3. Secondary Outcome: Change From Baseline to 12 Weeks, Benign Prostatic Hyperplasia (BPH) Impact Index
Description: The BII is a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores range from 0 to 13; higher scores represent increased perceived impact of benign prostatic hyperplasia-lower urinary tract symptoms on overall health. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population includes all subjects who were randomized, started study medication, and had non-missing data at baseline and Week 12. For the 12 week analysis, the LOCF imputation technique was used.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 163
Units on a Scale | -1.8 (0.21) | -1.3 (0.21)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.057, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for BII. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.6, Standard Error of Mean 0.3

4. Secondary Outcome: Change From Baseline to 12 Weeks, International Prostate Symptom Score (IPSS) Storage (Irritative) Subscore
Description: IPSS irritative subscore is the sum of Questions 2, 4 and 7 of the IPSS questionnaire. Scores range from 0 (few irritative symptoms) to 5 (frequent irritative symptoms), thus the 3 questions of the irritative subscore range from 0 to 15. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population was defined as all randomized subjects who started study medication, and had non-missing data at baseline and at least one post-baseline measurement. The LOCF imputation technique was employed.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 164
Units on a Scale | -2.3 (0.22) | -1.3 (0.21)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.002, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IPSS storage subscore. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.30

5. Secondary Outcome: Change From Baseline to 12 Weeks, International Prostate Symptom Score (IPSS) Voiding (Obstructive) Subscore
Description: IPSS obstructive subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 0 (few obstructive symptoms) to 5 (frequent obstructive symptoms), thus the 4 questions of the obstructive score range from 0 to 20. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 164
Units on a Scale | -3.3 (0.31) | -2.3 (0.31)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.020, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IPSS voiding subscore. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -1.0, Standard Error of Mean 0.43

6. Secondary Outcome: Change From Baseline to 12 Weeks, International Prostate Symptom Score (IPSS) Nocturia Question
Description: Measures nocturia (the need to get up at night to urinate). Scores range from 0 (few episodes of nocturia) to 5 (frequent episodes of nocturia). LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 164
Units on a Scale | -0.5 (0.08) | -0.4 (0.08)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.233, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IPSS nocturia question. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.1, Standard Error of Mean 0.11

7. Secondary Outcome: Change From Baseline to 12 Weeks, International Prostate Symptom Score (IPSS) Quality of Life (QoL) Index
Description: Assessment of QoL by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible). LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 160 | 164
Units on a Scale | -1.0 (0.10) | -0.7 (0.10)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.013, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IPSS QoL Index. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.4, Standard Error of Mean 0.15

8. Secondary Outcome: Patient Global Impression of Improvement (PGI-I), Number of Participants in 7 Response Categories
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: 12 weeks
Population: The analysis population includes all subjects who were randomized, started study medication, and had non-missing data.
Measure: Number; unit: Participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 155 | 158
Participants
  7-Very Much Worse | 1 | 0
  6-Much Worse | 5 | 6
  5-A Little Worse | 4 | 4
  4-No Change | 30 | 57
  3-A Little Better | 57 | 53
  2-Much Better | 46 | 32
  1-Very Much Better | 12 | 6
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — The p-value associates with difference between treatment groups for the 7 response categories; Results were adjusted for baseline LUTS severity (moderate [total IPSS < 20]; severe [total IPSS >= 20]

9. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I), Number of Participants in 7 Response Categories
Description: Measures clinician's perception of patient improvement at the time of assessment compared with the start of treatment. Scores range from 1 (very much better) to 7 (very much worse).
Time Frame: 12 weeks
Population: All values are based on the number of subjects in the analysis population with non-missing data.
Measure: Number; unit: Participants
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 155 | 158
Participants
  7-Very Much Worse | 0 | 0
  6-Much Worse | 5 | 2
  5-A Little Worse | 4 | 10
  4-No Change | 36 | 59
  3-A Little Better | 58 | 55
  2-Much Better | 39 | 25
  1-Very Much Better | 13 | 7
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — The p-value associates with difference between treatment groups for the 7 response categories; Results were adjusted for baseline LUTS severity (moderate [total IPSS < 20]; severe [total IPSS >= 20]

10. Secondary Outcome: Change From Baseline to 1 Week, International Prostate Symptom Score (IPSS)
Description: The IPSS Total Score is obtained by combining the scores of the responses to Question 1 through Question 7. Each question is scored from 0-5 for a total IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 1 week
Population: The analysis population includes all subjects who were randomized, started study medication, and had non-missing data at baseline and Week 1.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 147 | 150
Units on a Scale | -3.4 (0.35) | -2.7 (0.35)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.146, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 1 week between treatment groups for IPSS. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -0.7, Standard Error of Mean 0.49

11. Secondary Outcome: Change From Baseline to 4 Weeks, International Prostate Symptom Score (IPSS)
Description: as for outcome 10
Time Frame: Baseline, 4 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 158 | 162
Units on a Scale | -5.3 (0.43) | -3.5 (0.43)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 4 weeks between treatment groups for IPSS. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = -1.8, Standard Error of Mean 0.60

12. Secondary Outcome: Change From Baseline to 12 Weeks, International Index of Erectile Function (IIEF)- Erectile Function (EF) Domain Scores
Description: Self-reported EF. Scores range from 0 (low or no EF) to 5 (high EF) on 6 questions (1-5, 15 of the IIEF). EF Domain scores range from 0 to 30. LS mean of change from baseline to endpoint is from an ANCOVA. The model includes terms for treatment group, region, centered-baseline covariate, centered-baseline-by-treatment interaction and treatment-by-region interaction.
Time Frame: Baseline, 12 weeks
Population: The analysis population was defined as all randomized subjects who started study medication, and had non-missing data at baseline and at least one post-baseline measurement. Measures were taken only for those subjects who reported they were sexually active and reported erectile dysfunction. The LOCF imputation technique was employed.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 88 | 84
Units on a Scale | 6.7 (0.80) | 2.0 (0.82)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA — The p-value associates with LS Mean difference of changes from baseline to 12 weeks between treatment groups for IIEF-EF domain score. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment; Mean Difference (Final Values) = 4.7, Standard Error of Mean 1.12

13. Secondary Outcome: Change From Baseline to 12 Weeks, Peak Flow Rate (Qmax) by Uroflowmetry
Description: Qmax was defined as the peak urine flow rate (measured in milliliters per second [mL/sec] using standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 milliliters (mL) and the voided volume (Vcomp) was >=125 mL.
Time Frame: Baseline, 12 weeks
Population: The analysis population was defined as all randomized subjects who started study medication, and had non-missing data at baseline and at endpoint (considered the last non-missing post-baseline value).
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 127 | 135
mL/sec | 1.6 (4.64) | 1.1 (4.64)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.300, ranked ANOVA — The p-value associates with mean difference of changes from baseline to 12 weeks between treatment groups for Qmax. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment

14. Secondary Outcome: Change From Baseline to 12 Weeks, Mean Flow Rate (Qmean) by Uroflowmetry
Description: Qmean was defined as the mean urine flow rate (measured in mL/sec using standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 mL and the Vcomp was >=125 mL.
Time Frame: Baseline, 12 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 127 | 135
mL/sec | 0.6 (2.93) | 0.5 (2.79)

15. Secondary Outcome: Change From Baseline to 12 Weeks, Voided Volume (Vcomp) by Uroflowmetry
Description: Vcomp was defined as the volume of urine voided (measured in mL using standard calibrated flowmeter). At each visit, a uroflowmetry assessment was considered valid and the data were included in the statistical analyses only if the prevoid total bladder volume (assessed by ultrasound) was >=150 to <=550 mL and the Vcomp was >=125 mL.
Time Frame: Baseline, 12 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 127 | 135
mL | 16.9 (88.74) | 3.9 (105.68)

16. Secondary Outcome: Change From Baseline to 12 Weeks, Postvoid Residual (PVR) Volume
Description: The amount of urine remaining in the bladder after void completion.
Time Frame: Baseline, 12 weeks
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 154 | 158
mL | 8.8 (56.40) | 4.5 (66.71)
Statistical Analysis 1: Comparison: Tadalafil vs Placebo; Test type: Superiority or Other; p = 0.500, ranked ANOVA — The p-value associates with mean difference of changes from baseline to 12 weeks between treatment groups for PVR volume. Under the pre-specified fixed sequence testing procedure, the significance level of 0.05 is used for assessment

ADVERSE EVENTS:
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 2/161 | 0/164
Other Adverse Events (participants affected / at risk) | 41/161 | 36/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=161) | Placebo (N=164)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — This event resulted in death.
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=161) | Placebo (N=164)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (2) | 1 (2)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (4)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vertebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endoscopy (Investigations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days